CLINICAL TRIAL: NCT06886048
Title: Effects of Barley Green on Visceral Fat Area in the Human Body and Investigation Into the Associated Mechanism of Intestinal Microbiota
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Cui Mingxuan, Principal Investigator, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024PHB574-001
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: People With High Body Fat Percentage; People With High Visceral Fat Area

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (No Intervention)
- intervention group (Experimental)
  Interventions: Dietary Supplement: barley green

INTERVENTIONS:
Dietary Supplement: barley green — Oral administration: 30 minutes before meals Dosage: 4 g powder, 5 g tablet Frequency: 2 times a day
  Arms: intervention group

SUMMARY:
The aim of this study was to investigate the changes in visceral fat area and associated indicators in individuals with high body fat percentage under the intervention of barley green, elucidate the clinical efficacy of barley green on human visceral fat, and preliminarily explore the mechanism by which barley green influences human visceral fat through gut microbiota analysis. Participants with high body fat percentage were recruited from the Clinical Nutrition Department of Peking University People's Hospital and randomly assigned to either an intervention group or a control group. The intervention group received a regimen combining barley green supplementation with a calorie-restricted balanced diet plan, while the control group followed only the calorie-restricted balanced diet plan. General clinical data were collected, nutritional assessments were conducted, and dynamic analyses of body composition and metabolism were performed. Venous blood samples were obtained for the measurement of metabolic and inflammation-related indices as well as gut microbiota characterization. By observing and comparing differences in visceral fat area and related parameters, as well as gut microbiota profiles between the two groups, this study provides a scientific foundation for the clinical application of barley green in medical nutrition interventions targeting populations with high body fat percentage.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years old, gender is not limited; Body fat percentage exceeding the upper limit of the standard range: male > 20%, female > 28%; Visceral fat area > 100cm2; Willing to accept the assessment and sign informed consent.

Exclusion Criteria:

* ① Patients currently receiving weight-loss medications (e.g., incretin-based therapies such as GLP-1 receptor agonists) or medications that improve insulin resistance (e.g., metformin or other insulin-sensitizing agents), or anti-inflammatory agents with documented effects on inflammatory markers (including but not limited to lipid-lowering agents, hypoglycemic agents, antihypertensives, urate-lowering agents, etc.);

  * Patients concurrently using nutritional supplements or functional foods (e.g., phytochemicals, health supplements) with demonstrated effects on reducing body fat or visceral adiposity;

    * Patients regularly consuming prebiotics, probiotics, or other microbiota-modulating agents;

      * Patients with diseases severely affecting nutrient digestion or absorption (e.g., chronic diarrhea, severe constipation, active inflammatory bowel disease, active gastrointestinal ulcers, history of gastrointestinal resection, cholecystitis/post-cholecystectomy syndrome, etc.);

        * Patients with cardiovascular/cerebrovascular diseases (e.g., coronary artery disease, heart failure, arrhythmias, cardiomyopathies, cerebral infarction, cerebral hemorrhage, cerebral arteritis), grade 3 hypertension, stroke, chronic hepatitis, malignancies, anemia, psychiatric disorders, cognitive impairment, epilepsy, acute-phase gout, nephrolithiasis, or renal insufficiency;

          ⑥ Patients with hepatic dysfunction (alanine aminotransferase [ALT] and/or aspartate aminotransferase [AST] levels exceeding 3 times the upper limit of normal [ULN]) or renal dysfunction (serum creatinine exceeding ULN);

          ⑦ Patients with active infectious diseases (e.g., tuberculosis, HIV/AIDS);

          ⑧ Patients with severe allergies to any component of the investigational products;

          ⑨ Pregnant or lactating individuals;

          ⑩ Patients with physical disabilities or other conditions deemed ineligible by investigators (e.g., clinically significant comorbidities not listed above).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
visceral fat area in cm2 | From enrollment to the end of treatment at 8 weeks.
  Visceral fat areas are measured by the Inbody 770 instrument at two time points: the day of enrollment and 8 weeks after enrollment.

SECONDARY OUTCOMES:
height in centimeters | From enrollment to the end of treatment at 8 weeks
  Height in centimeters are measured by Manual Height Ruler at two time points: the day of enrollment and 8 weeks after enrollment.
weight in kilograms | From enrollment to the end of treatment at 8 weeks
  Weight in kilograms are measured by the Inbody 770 instrument at two time points: the day of enrollment and 8 weeks after enrollment.
BMI in kg/m^2 | From enrollment to the end of treatment at 8 weeks
  Weight and height will be combined to report BMI in kg/m^2 at two time points: the day of enrollment and 8 weeks after enrollment.
body fat rate in % | From enrollment to the end of treatment at 8 weeks
  Body fat rates are measured by the Inbody 770 instrument at two time points: the day of enrollment and 8 weeks after enrollment.
muscle mass in kilograms | From enrollment to the end of treatment at 8 weeks
  Muscle masses are measured by the Inbody 770 instrument at two time points: the day of enrollment and 8 weeks after enrollment.
basal metabolic rate in kcal | From enrollment to the end of treatment at 8 weeks
  Basal metabolic rates are measured by the Inbody 770 instrument at two time points: the day of enrollment and 8 weeks after enrollment.
skeletal muscle mass in kilograms | From enrollment to the end of treatment at 8 weeks
  Skeletal muscle masses are measured by the Inbody 770 instrument at two time points: the day of enrollment and 8 weeks after enrollment.
blood pressure in mmHg | From enrollment to the end of treatment at 8 weeks
  Blood pressures are measured by electronic blood pressure monitor at two time points: the day of enrollment and 8 weeks after enrollment.
waist circumference in millimeters | From enrollment to the end of treatment at 8 weeks
  Waist circumferences are measured by tape measure at two time points: the day of enrollment and 8 weeks after enrollment.
hip circumference in millimeters | From enrollment to the end of treatment at 8 weeks
  Hip circumferences are measured by tape measure at two time points: the day of enrollment and 8 weeks after enrollment.
upper arm circumference in millimeters | From enrollment to the end of treatment at 8 weeks
  Upper arm circumferences are measured by tape measure at two time points: the day of enrollment and 8 weeks after enrollment.
left hand grip strength in pound-force | From enrollment to the end of treatment at 8 weeks
  Left hand grip strengths are measured by grip dynamometer at two time points: the day of enrollment and 8 weeks after enrollment.
right hand grip strength in pound-force | From enrollment to the end of treatment at 8 weeks
  Right hand grip strengths are measured by grip dynamometer at two time points: the day of enrollment and 8 weeks after enrollment.
triceps skinfold thickness in millimeters | From enrollment to the end of treatment at 8 weeks
  Triceps skinfold thicknesses are measured by skin fold thickness gauge at two time points: the day of enrollment and 8 weeks after enrollment.
subscapular horn skinfold thickness in millimeters | From enrollment to the end of treatment at 8 weeks
  Subscapular horn skinfold thicknesses are measured by skin fold thickness gauge at two time points: the day of enrollment and 8 weeks after enrollment.
abdominal skinfold thickness in millimeters | From enrollment to the end of treatment at 8 weeks
  Abdominal skinfold thicknesses are measured by skin fold thickness gauge at two time points: the day of enrollment and 8 weeks after enrollment.
food intake dose in grams | From enrollment to the end of treatment at 8 weeks
  Data of food intake doses are taken by food frequency questionnaire and 3-day food diary at two time points: the day of enrollment and 8 weeks after enrollment.
uric acid levels in umol/L | From enrollment to the end of treatment at 8 weeks
  Uric acid levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
blood glucose in mmol/L | From enrollment to the end of treatment at 8 weeks
  Blood glucose levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
total cholesterol in mmol/L | From enrollment to the end of treatment at 8 weeks
  Total cholesterol levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
triglycerides in mmol/L | From enrollment to the end of treatment at 8 weeks
  Triglycerides levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
high-density lipoprotein cholesterol in mmol/L | From enrollment to the end of treatment at 8 weeks
  High-density lipoprotein cholesterol levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
low-density lipoprotein cholesterol in mmol/L | From enrollment to the end of treatment at 8 weeks
  Low-density lipoprotein cholesterol levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
white blood cell count in 10^9/L | From enrollment to the end of treatment at 8 weeks
  White blood cell counts are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
hemoglobin in g/L | From enrollment to the end of treatment at 8 weeks
  Hemoglobin levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
glutamic-pyruvic transaminase in U/L | From enrollment to the end of treatment at 8 weeks
  Glutamic-pyruvic transaminase levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
glutamic oxalacetic transaminase in U/L | From enrollment to the end of treatment at 8 weeks
  Glutamic oxalacetic transaminase levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
albumin in g/L | From enrollment to the end of treatment at 8 weeks
  Albumin levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
vitamin B6 in ng/mL | From enrollment to the end of treatment at 8 weeks
  Vitamin B6 levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
vitamin B1 in ng/mL | From enrollment to the end of treatment at 8 weeks
  Vitamin B1 levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
vitamin B9 in ng/mL | From enrollment to the end of treatment at 8 weeks
  Vitamin B9 levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
vitamin B5 in ng/mL | From enrollment to the end of treatment at 8 weeks
  Vitamin B5 levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
vitamin B3 in ng/mL | From enrollment to the end of treatment at 8 weeks
  Vitamin B3 levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
vitamin B2 in ng/mL | From enrollment to the end of treatment at 8 weeks
  Vitamin B2 levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
vitamin B12 in ng/mL | From enrollment to the end of treatment at 8 weeks
  Vitamin B12 levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
vitamin A in ng/mL | From enrollment to the end of treatment at 8 weeks
  Vitamin A levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
vitamin D in ng/mL | From enrollment to the end of treatment at 8 weeks
  Vitamin D levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
vitamin E in ng/mL | From enrollment to the end of treatment at 8 weeks
  Vitamin E levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
vitamin K in ng/mL | From enrollment to the end of treatment at 8 weeks
  Vitamin K levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
cobalt in µg/L | From enrollment to the end of treatment at 8 weeks
  Cobalt levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
nickel in µg/L | From enrollment to the end of treatment at 8 weeks
  Nickel levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
selenium in µg/L | From enrollment to the end of treatment at 8 weeks
  Selenium levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
arsenic in µg/L | From enrollment to the end of treatment at 8 weeks
  Arsenic levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
platinum in µg/L | From enrollment to the end of treatment at 8 weeks
  Platinum levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
copper in mg/L | From enrollment to the end of treatment at 8 weeks
  Copper levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
molybdenum in µg/L | From enrollment to the end of treatment at 8 weeks
  Molybdenum levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
zinc in mg/L | From enrollment to the end of treatment at 8 weeks
  Zinc levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
manganese in µg/L | From enrollment to the end of treatment at 8 weeks
  Manganese levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
magnesium in mg/L | From enrollment to the end of treatment at 8 weeks
  Magnesium levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
cadmium in µg/L | From enrollment to the end of treatment at 8 weeks
  Cadmium levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
iron in mg/L | From enrollment to the end of treatment at 8 weeks
  Iron levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
thallium in µg/L | From enrollment to the end of treatment at 8 weeks
  Thallium levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
lead in µg/L | From enrollment to the end of treatment at 8 weeks
  Lead levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
calcium in mg/L | From enrollment to the end of treatment at 8 weeks
  Calcium levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
cortisol in µg/dL | From enrollment to the end of treatment at 8 weeks
  Cortisol levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
growth hormone in ng/mL | From enrollment to the end of treatment at 8 weeks
  Growth hormone levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
fasting insulin in uU/mL | From enrollment to the end of treatment at 8 weeks
  Fasting insulin levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
thyroid-stimulating hormone in uIU/mL | From enrollment to the end of treatment at 8 weeks
  Thyroid-stimulating hormone levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
free thyroxine in pmol/L | From enrollment to the end of treatment at 8 weeks
  Free thyroxine levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
free triiodothyronine in pmol/L | From enrollment to the end of treatment at 8 weeks
  Free triiodothyronine levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
IL-1β in pg/mL | From enrollment to the end of treatment at 8 weeks
  IL-1β levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
IL-6 in pg/mL | From enrollment to the end of treatment at 8 weeks
  IL-6 levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
IL-10 in pg/mL | From enrollment to the end of treatment at 8 weeks
  IL-10 levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
leptin in pg/mL | From enrollment to the end of treatment at 8 weeks
  Leptin levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
adiponectin in µg/mL | From enrollment to the end of treatment at 8 weeks
  Adiponectin levels are measured by blood samples at two time points: the day of enrollment and 8 weeks after enrollment.
Hardness of liver in kPa | From enrollment to the end of treatment at 8 weeks
  Hardness of liver is measured by Liver Ultrasound Elastography at two time points: the day of enrollment and 8 weeks after enrollment.
Controlled Attenuation Parameter in dB/m | From enrollment to the end of treatment at 8 weeks
  Controlled Attenuation Parameter is measured by Liver Ultrasound Elastography at two time points: the day of enrollment and 8 weeks after enrollment.
Alpha diversity (Shannon index, Chao1) | From enrollment to the end of treatment at 8 weeks
  Alpha diversity is measured by fecal specimen assessed by 16S rRNA sequencing at two time points: the day of enrollment and 8 weeks after enrollment.
Beta diversity (Bray-Curtis dissimilarity) | From enrollment to the end of treatment at 8 weeks
  Beta diversity is measured by fecal specimen assessed by 16S rRNA sequencing at two time points: the day of enrollment and 8 weeks after enrollment.
Relative abundance of specific taxa (e.g., Firmicutes/Bacteroidetes ratio) | From enrollment to the end of treatment at 8 weeks
  Relative abundance of specific taxa is measured by fecal specimen assessed by 16S rRNA sequencing at two time points: the day of enrollment and 8 weeks after enrollment.
Predicted functional pathways (via metagenomic analysis) | From enrollment to the end of treatment at 8 weeks
  Predicted functional pathways are analyzed via metagenomic analysis after 16S rRNA sequencing at two time points: the day of enrollment and 8 weeks after enrollment.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Xicheng District, China

IPD SHARING:
Plan to Share IPD: Undecided